CLINICAL TRIAL: NCT01657201
Title: A Randomized, Open-label, Two-Treatment, Two-Period, Two-Sequence, Cross-over Study to Evaluate the Pharmacokinetic Properties of SYP-1018 (Voriconazole-loaded PNP) and Voriconazole (Vfend) in Healthy Male Volunteers
Brief Title: Study to Evaluate the Pharmacokinetic Properties of SYP-1018 (Voriconazole-loaded PNP) and Voriconazole (Vfend)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SYP1018
Record Dates: First submitted 2012-07-29; First posted 2012-08-06 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Systemic Mycotic Infection
MeSH Terms: interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): SYP-1018 200mg → Voriconazole 200mg
  Interventions: Drug: SYP-1018 200mg; Drug: Voriconazole 200mg
- Sequence 2 (Experimental): Voriconazole 200mg → SYP-1018 200mg
  Interventions: Drug: SYP-1018 200mg; Drug: Voriconazole 200mg

INTERVENTIONS:
Drug: SYP-1018 200mg — SYP-1018 200mg, Intravenous administration
Drug: Voriconazole 200mg — Voriconazole 200mg, Intravenous administration

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic properties and safety of SYP-1018 (Voriconazole-loaded PNP) and Voriconazole (Vfend).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 20-45 years of age
* Weight of ≥ 60kg ≤ 90kg with BMI of ≥ 19 and < 27 (BMI(kg/m2)= weight(kg)/{height(m)}2
* Voluntary written informed consent

Exclusion Criteria:

* History or presence of significant renal, neurologic, pulmonary, endocrine, hematology, oncology, urologic, cardiovascular, musculoskeletal or psychiatric disease
* Drug allergies to Voriconazole
* Recent history or evidence of drug abuse
* Recent participation(within 2 months) in other clinical studies
* Recent donation of blood(within 2months), plasma(within 1month) or transfusion(within 1month)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters | pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24h
  AUClast, Cmax

SECONDARY OUTCOMES:
Pharmacokinetics parameters | pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24h
  AUCinf, Tmax, T1/2, CL
Safety | 16 days
  Adverse events, Laboratory assessments, Vital signs, Electrocardiograms(ECGs)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Institute, Seoul National University Hospital, Seoul, South Korea